CLINICAL TRIAL: NCT06681090
Title: Effectiveness of Low-Level Laser Therapy and Topical Steroid Therapy in the Management of Oral Lichen Planus
Brief Title: Different Treatment Modalities for Oral Lichen Plan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Asem Mohammed Kamel Ali, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Management of Oral Lichen Plan
Record Dates: First submitted 2024-11-02; First posted 2024-11-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Oral Lichen Planus
Keywords: Low-Level Laser; Topical Steroid; 0.1% triamcinolone acetonide; management of oral lichen planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Out of all the researchers, only one had knowledge of the patients' assigned groups. Neither the therapies nor their efficacy was evaluated by this unblinded researcher. There was a lack of treatment blinding for patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Steroid Therapy of Erosive oral lichen planus (Experimental): topical application of 0.1% triamcinolone acetonide and photo biomodulation on erosive oral lichen planus, 3 times daily and a miconazole oral gel once daily, for 4 weeks
  Interventions: Drug: 0.1% topical triamcinolone Acetonide preparation "Kenacourt-A Orabase"
- Low-Level Laser Therapy of Erosive oral lichen planus (Experimental): Photo biomodulation with laser therapy twice a week for 8 sessions over 4 weeks, utilizing a 980 nm diode laser with an output power of 300 mw.
  Interventions: Device: 980 nm diode laser

INTERVENTIONS:
Drug: 0.1% topical triamcinolone Acetonide preparation "Kenacourt-A Orabase" — The patients were administered topical corticosteroids in the form of a 0.1% triamcinolone acetonide preparation (Kenacort TM 0.1% Abbott). The medication was to be used 3 times every day for 4 weeks or until the lesion has healed, whichever occurs first. After applying the gel, the patients were instructed not to consume any fluids or food for at least 1 hour. In addition, a topical antifungal treatment consisting of Miconazole oral gel at a concentration of 2% should be applied once a day for 4 weeks
  Arms: Topical Steroid Therapy of Erosive oral lichen planus
Device: 980 nm diode laser — First group (Group A) underwent PBM therapy using a 980 nm diode laser (elexxion nano dental laser with a flat top handpiece). The therapy included 8 sessions for 4 weeks, with 2 sessions conducted per week, all administered by the same operator. The energy was evenly distributed across all the mucosal lesions and the surrounding tissues within a 0.5 cm range using a spot-technique method with little overlap.
  Arms: Low-Level Laser Therapy of Erosive oral lichen planus

SUMMARY:
The goal of applications of Low-Level Laser and Topical Steroid in the Management of Oral Lichen Planus is to learn if intervention can by relieve pain, decreasing inflammation, and facilitating tissue healing in20 patients who were suffering from erosive oral lichen planus. The main questions it aims to answer are which is better and more effective as treatment modality. The erosion size (mm2) measured on the first day and 4 weeks later. Oral Health-Related Quality of Life questionnaire manipulated. Researchers will take Low-Level Laser and Topical Steroid in the Management of Oral Lichen Planus to see if it could be used as separate treatment option or as combination.

ELIGIBILITY:
Inclusion Criteria:

* patients who were monitored for OLP.
* clinical and histopathological finding of OLP in accordance with van der Meij 2003.
* being over 18 years old.

Exclusion Criteria:

* Patients with systemic disorders, pregnancy, using drugs, smoking, lesions in contact with dental amalgams, and cutaneous or other mucosal involvement at the time of treatment were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
The erosion size | From enrollment to the end of treatment at 4 weeks"
  The maximal diameter (mm) and width (mm) were measured perpendicularly using a calibrated periodontal probe
The Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 4 weeks"
  pain ratings span from zero (indicating the absence of pain) to 10 (representing extremely intense pain) along a horizontal line values. { the minimum is 0 and maximum is 10 }

SECONDARY OUTCOMES:
Oral Health-Related Quality of Life (OHRQoL) | From enrollment to the end of treatment at 4 weeks"
  A month following the initial appointment, participants were asked about the OLP that had restricted their everyday activities. The 8 tasks included eating, talking, cleaning one's mouth, sleeping, smiling, laughing freely, maintaining emotional stability, performing strenuous physical labour, and interacting with others. { the minimum is 0 and maximum values is 5 }.a score of zero indicated never being afflicted, a score of 1 meant once a month, a score of 2 meant twice a month, scoring 3 indicated a frequency of once or twice weekly, 4 indicated 3 to 4 times weekly, and 5 signified daily or very daily occurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F. Assistant Professor, PhD, Principal Investigator — Faculty of Dentistry, Assiut University, Egypt; Rahma M. Lecturer, PhD, Principal Investigator — Faculty of Dentistry, Assiut University, Egypt; Asem K. Lecturer, PhD, Study Chair — Dental Medicine Faculty, Al-Azhar University (Assiut Branch), Assiut, Egypt; Mahmoud A. Professor, PhD, Study Director — Faculty of Dentistry, Al-Azhar University (Assiut Branch), Assiut, Egypt.
Locations (1):
- Faculty of Dentistry, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Meij EH, Schepman KP, van der Waal I. The possible premalignant character of oral lichen planus and oral lichenoid lesions: a prospective study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Aug;96(2):164-71. doi: 10.1016/s1079-2104(03)00305-6. PMID 12931088
- [Background] Ruiz Roca JA, Lopez Jornet P, Gomez Garcia FJ, Marcos Aroca P. Effect of Photobiomodulation on Atrophic-Erosive Clinical Forms of Oral Lichen Planus: A Systematic Review. Dent J (Basel). 2022 Nov 27;10(12):221. doi: 10.3390/dj10120221. PMID 36547037
- [Background] Bhatt G, Gupta S, Ghosh S. Comparative efficacy of topical aloe vera and low-level laser therapy in the management of oral lichen planus: a randomized clinical trial. Lasers Med Sci. 2022 Apr;37(3):2063-2070. doi: 10.1007/s10103-021-03480-1. Epub 2021 Dec 1. PMID 34853932